CLINICAL TRIAL: NCT03441009
Title: Metabolism and the Activity of the Autonomic Nervous System in Patients With Paroxystic Sympathetic Hyperactivity, PSH
Acronym: MANS-PSH
Status: Completed | Type: Observational
Sponsor: Region MidtJylland Denmark (Other)
Responsible Party: Principal Investigator, Soren Sondergaard, Senior Consultant, Region MidtJylland Denmark
Other Study IDs: 654865
Record Dates: First submitted 2018-02-09; First posted 2018-02-22 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Autonomic Nervous System Imbalance
Keywords: PSH, Rehabilitation, Medication, ANS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Physio-/occupational therapy — Physio-/occupational therapy, ADL
  Other Names: Psycotropic medications

SUMMARY:
Adult patients suffering from acquired brain damage run the risk of developing PSH. This group of patients is admitted to our unit, the Neurointensive Stepdown Unit, at Silkeborg Regional Hospital for intensive care and early neurorehabilitation. After weaning from intensive carethey are transferred to Hammel NeuroCentre.

Aim is to assess whether HRV-derived variables in the frequency domain mirror therapeutic and/or nursing and/or pharmacologic interventions. To the extent clinically available BRS and metabolism are included in the assessment.

DETAILED DESCRIPTION:
See report:

Honore H, Eggertsen K, Sondergaard S: A study into the feasibility of using HRV variables to guide treatment in patients with paroxystic sympathetic hyperactivity in a neurointensive step-down unit. NeuroRehabilitation 2019, 44(1):141-155.

ELIGIBILITY:
Inclusion Criteria:

Symptoms of PSH according to Baguley scoring table

Exclusion Criteria:

No symptoms of PSH

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to NISU from tertiary health care facilities for intensive care in combination with early neurorehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Difference before vs after intervention in frequency domain parameters of HRV | immediate
  HRV parameters: low frequency (LF, 0.04-0.15 Hz), high frequency (HF, 0.15-0.4 Hz) in terms of peak frequency (Hz), absolute power (ms2, natural logarithm transformed values of absolute powers of VLF, LF, and HF bands), relative power (absolute power/total power), normalized power (%, normalized units, n.u.), total power given by VLF + HF + LF (ms2) and LF/HF ratio.
Qualitative description expressed as goal attainment scaling (GAS) of therapeutic interventions | immediate
  Two independent ratings on a 5-point scale, -2 to +2

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen Feldbæk, Professor, Study Chair — Hammel Neuro- and Research Centre

IPD SHARING:
Plan to Share IPD: No